CLINICAL TRIAL: NCT04063865
Title: Protection of Renal Function After Liver Transplant Using Everolimus Monotherapy as the Immunosuppression Regimen
Brief Title: Everolimus Monotherapy as Immunosuppression After Liver Transplant
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was larger than expected and became a burden to faculty and staff resources.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Chandrashekhar Kubal, Princial Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1807401376
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Results first posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Tacrolimus; Everolimus

STUDY DESIGN:
Intervention Model Description: Tacrolimus as maintenance immunosuppression
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Arm (Active Comparator): Tacrolimus as maintenance immunosuppression
  Interventions: Drug: Tacrolimus
- Study Arm (Experimental): Everolimus monotherapy maintenance immunosuppression
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus (FK / Prograf) titrated to a goal trough of 6 - 8 ng/ml
  Other Names: Prograf
  Arms: Control Arm
Drug: Everolimus — Everolimus monotherapy - target trough levels 4 - 8 ng/ml as maintenance immunosuppression
  Other Names: Zortress
  Arms: Study Arm

SUMMARY:
Tacrolimus is the standard immunosuppressive drug used to prevent organ rejection post liver transplant. One side effect of Tacrolimus is nephrotoxicity. Everolimus does not have the nephrotoxicity side effects of Tacrolimus.

Replacement of Tacrolimus by Everolimus may have a reduced incidence of renal dysfunction in liver transplant patients who have near normal kidney function prior to liver transplantation. Other investigators have already shown a benefit in terms of renal function with introduction of Everolimus with reduced-exposure tacrolimus at 1 month after liver transplantation, this benefit has been shown was maintained to 3 years in patients who continued Everolimus therapy with comparable efficacy and no late safety concerns. Investigators in this trial are proposing to advance this approach further by completely eliminating Tacrolimus from patients' immunosuppression protocol. The rationale for this approach is based on a unique induction immunosuppression protocol.

Liver transplant patients receive potent induction immunosuppression in the form of rabbit anti thymocyte globulin.

Investigators believe that in conjunction with this induction regimen, patients can be maintained on Everolimus monotherapy without the risk of rejection. By completely eliminating Tacrolimus, investigators believe that there may be further benefit in terms of renal function. Additionally, Everolimus is known to induce tolerance in transplant recipients. Tolerant patients do not require immunosuppression to accept transplant organs.

The long-term efficacy and safety of Everolimus monotherapy as the maintenance immunosuppression in patients receiving rATG induction is unknown.

Primary Aim: Assess the effect of Everolimus monotherapy versus Tacrolimus monotherapy on long term renal function measured by Glomerular Filtration Rate (GFR).

DETAILED DESCRIPTION:
Following enrollment, subjects will be randomized at one month post transplant to Tacrolimus (control) or to Everolimus (study) as maintenance immunosuppression.

After liver transplant, all patients will receive the standard induction regimen and Tacrolimus monotherapy.

INDUCTION:

Rabbit anti-thymocyte globulin (rATG) 1.5 mg/kg of actual body weight rounded to nearest 25 mg and capped at 150 mg for up to three doses given IV on post-operative day (POD) 1, 3, and 5. Some patients may receive only one dose if considered too frail to need all three doses.

30 minutes prior to infusion, pre-medicate with the following: Daily steroid dose Acetaminophen (Tylenol®) 650 mg PO or per nasogastric (NG) x 1 dose Diphenhydramine (Benadryl®) 25 mg IV push x 1 dose

Steroids:

Methylprednisolone (Solu-Medrol®) 250 mg IV push x 1 dose on POD 1 (given 30 minutes prior to rATG) and 125 mg IV push x 1 dose on POD 3.

Maintenance:

Tacrolimus (FK / Prograf®) (titrated to a goal trough of 6 - 8 ng/mL).

RANDOMIZATION:

On POD 30, patients meeting study criteria will be randomized to either the study arm or control arm. Patients randomized to the study arm will be converted to Everolimus (target trough levels 4 - 8 ng/mL) + low dose Tacrolimus (target trough levels 3-5 ng/mL) (study arm). The control arm will be maintained on the Tacrolimus monotherapy (target trough levels 6-8 ng/mL).

At 3 months, patients in the study arm will be gradually weaned off of Tacrolimus over a period of one month to remain on Everolimus monotherapy (target trough levels 4-8 ng/mL). Patients in the control arm will remain on tacrolimus monotherapy (target trough levels 6-8 ng/mL).

Complete blood counts, liver function panels, and drug levels will be monitored as done Standard of Care [SOC]:

initially twice per week for first month, once per week for next two months, once every other week for next three weeks, and then once monthly. Ultrasound, endoscopic retrograde cholangiopancreatography (ERCP), biopsy as needed by clinical situation as SOC.

For characterizing operational tolerance in these patients, investigators will use a 13#gene set to predict liver transplant tolerance has been identified and validated by others.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant recipients >= 18 years old
* Normal baseline renal dysfunction (GFR > 60 mL/min)
* Rabbit anti-thymocyte globulin (rATG) induction (cumulative dose 1.5 - 5 mg/kg)
* Indication for transplant: ethanol, hepatitis C, or nonalcoholic steatohepatitis or any combination of these

Exclusion Criteria:

* Increased risk of rejection: autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, positive crossmatch, retransplantation
* Incompletely healed incision or other wound healing issues at time of randomization
* Multiple or previous organ transplantation
* Severe, uncontrolled hypercholesterolemia (> 9mmol/L) or hypertriglyceridemia (>8.5 mmol/L) in the 6 months prior to transplantation
* Insurance company unwilling to pay for the cost of the everolimus or patient does not qualify for the Novartis Patient Assistance Program.
* Pregnant women
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandrashekhar Kubal, MD, Principal Investigator — Indiana University
Locations (1):
- IU Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Arm: Everolimus monotherapy maintenance immunosuppression
  Everolimus: Everolimus (target trough levels 4 - 8 ng/mL) + low dose Tacrolimus (target trough levels 3-5 ng/mL)
Period: Overall Study
Arm/Group | Control Arm | Study Arm
Started | 6 | 8
Completed | 0 | 0
Not Completed | 6 | 8
Not completed — Physician Decision | 1 | 3
Not completed — Study Closed Prior to Completion | 4 | 4
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Study Arm | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: Years] | 51.33 [48 to 59] | 57.5 [51 to 66] | 54.86 [48 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Long-Term Renal Function With Tacrolimus Monotherapy
Description: Glomerular Filtration Rate
Time Frame: 36 months post-transplant
Population: Study was terminated prior to any subject reaching the 36 Month timepoint. No data were collected for this outcome measure.
Arm/Group | Control Arm | Study Arm
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Long-Term Renal Function With Everolimus Monotherapy
Description: Glomerular Filtration Rate
Time Frame: 36 months post-transplant
Population: as for outcome 1
Arm/Group | Control Arm | Study Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year, 2 months
Description: AEs were collected from each participant for up to 14 months since the study was terminated prior to completion.
Arm/Group | Control Arm | Study Arm
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=6) | Study Arm (N=8)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — ED with chest pain and 3 days of fever. Chest x-ray showed left sided infiltrates and trace pleural effusion. Was started on IV antibiotics and fluids. Given Percocet for left sided chest wall pain. Did not stop Everolimus.
Liver Infection (Hepatobiliary disorders) | 1 (1) | 0 (0) — pt completed profylactic anti-viral therapy. First labs for CMV showed infection. He has been restarted on anti-virals. He was admitted for work up of elevated LFTs. He has had biopsy performed and is being treated for CMV currently.
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pt reported to ER for back pain. Was found on imaging and had thoracentesis performed. He returned and had this performed again on 5/19. Pt reports no further SoB as of 6/5/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT04063865/Prot_SAP_001.pdf